CLINICAL TRIAL: NCT04890665
Title: Effectiveness of a Self-applied Multi-component Psychological Online Intervention Based on User Experience, for Anxiety, Depression, Burnout, Fatigue Compassion on Healthcare Workers During the COVID-19 Outbreak: A Randomized Clinical Trial
Brief Title: Online Multi-component Psychological Intervention for Healthcare Workers During COVID-19 Pandemic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Internacional de Valencia (Other)
Collaborators: Universidad Autonoma de Ciudad Juarez (Other); University of Guadalajara (Other); Universidad Nacional Autonoma de Mexico (Other); Universidad Internacional del Ecuador (Other); University of Buenos Aires (Other); University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VIU-Health_care_workers_COVID
Record Dates: First submitted 2021-05-17; First posted 2021-05-18 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Anxiety; Depression; Sleep Disturbance; Quality of Life; Burnout, Professional; Stress; Fatigue, Compassion
MeSH Terms: conditions — Anxiety Disorders; Depression; Parasomnias; Burnout, Professional; Compassion Fatigue | interventions — Health Personnel

STUDY DESIGN:
Intervention Model Description: The study has two arms, one is the experimental group that receives the treatment solely through the online platform, and the other is the comparison group that will receive treatment delivered through a therapist through video calls. The patients in both groups will be evaluated pre and post/treatment. The participants are assigned randomly to the intervention or comparison group.
Who Masked: Participant
Masking Description: The patients are not aware that there is an experimental group and a control group, the participants are not related and do not know each other. The conditions of the study are only known by the researcher, the therapists, and the Research Ethics Committee of the Universidad Autónoma de Ciudad Juárez.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Self-applied psychological intervention for healthcare workers (Experimental): Participants in this group will receive 9 sessions of a multi-component psychological intervention focused on the reduction of symptoms of anxiety, depression, stress, burnout, fatigue compassion, and post-traumatic stress, and the increase of the quality of sleep and perception of the quality of life. The participants will have the option to do 3 extra modules that are complimentary for the intervention.
  Interventions: Behavioral: Online psychological intervention for healthcare workers
- Control: Self-applied psychological intervention for healthcare workers (Active Comparator): The participants in this group will receive exactly the same intervention but delivered through a therapist in a weekly session through an online video call. The participants will be informed also about the 3 extra modules and briefly what it is the contents of these modules so they can accept or not receive these extra contents.
  Interventions: Behavioral: Online psychological intervention for healthcare workers

INTERVENTIONS:
Behavioral: Online psychological intervention for healthcare workers — The intervention is based on Cognitive Behavioral Therapy, Mindfulness, Behavioral Activation Therapy, Acceptance and Commitment Therapy and Positive Psychology, aimed at the Psychoeducation regarding the manifestations of anxiety, depression, burnout, fatigue compassion, posttraumatic stress disorder, and affectations in sleep quality and perception of life quality in healthcare workers.
  And 3 complementary modules that according to the scientific literature could affect the mental health of healthcare workers related to how to deliver bad health news, Psychological first aid and how beliefs could influence physical and emotional self-care in the face of the COVID-19 pandemic.

SUMMARY:
The objective of this study is to carry out a randomized clinical trial with healthcare workers in Mexico through a web platform. The intervention aims to reduce anxiety, depressive symptoms, burnout, stress, compassion fatigue, and increase the quality of life and sleep and self-care, as well as improve skills in providing bad news to patients and their families. A self-applied intervention will be compared with an intervention delivered by therapists providing the same intervention implemented through Zoom, Skype, or Microsoft Teams, to ensure sanitary protection measures.

DETAILED DESCRIPTION:
Recent studies indicate that a lack of personal protective equipment, an unreasonable amount of work, inadequate medications, fear of contracting the disease, spreading the disease to co-workers and family, and lack of qualified training, have put front-line healthcare workers with unimaginable stress. There are various psycho social stressors to which the person who is working in this line of action is exposed. Nurses have been found to be one of the most affected groups because they have manifested various psychological consequences, including anxiety, depression, and stress. Likewise, multiple studies have reported psychological discomfort in health workers, especially those who are in areas of care for patients infected by COVID-19, among the most frequent psychological consequences that have been found, high prevalence of anxiety, depression, stress, insomnia, and high levels of distress are observed. Some of the challenges faced by health personnel who are in contact with patients infected by the virus are having a higher risk of contagion, not having the necessary personal equipment to prevent contagion, excessive workload, and even neglecting activities basic. In addition to these unfavorable working conditions faced by COVID-19 front line care staff, there is a need to make complex decisions that can generate moral or ethical damage. Consequently, this situation can trigger a series of negative emotional alterations, such as anxiety, depression, post-traumatic stress disorder, and even suicidal ideas.

Due to the current restrictions derived from the pandemic, psychological digital interventions have been an effective option to overcome barriers in mental health care for this population. Likewise, this type of intervention can provide various benefits, such as carried out by different means and the efficacy that they have shown to treat a wide range of mental health problems.

The objective of this study is to carry out a randomized clinical trial through a web platform which will have two groups: 1) Self-applied intervention directed at health personnel from all over Mexico for the reduction of symptoms of anxiety, depression, burnout, stress, compassion fatigue and increased self-care, quality of sleep and perceived quality of life, as well as how to offer tools to acquire knowledge about how to notify bad news to patients and families. The contents of the online intervention will be implemented through a responsive web application. In order to create the most fitted intervention for the real needs of the participants will be created following the principles of User Experience, this ensuring that the design characteristics of the tool will meet the desired requirements to be perceived as easy to use, attractive and useful. The User Experience approach refers to the experience that a user has with a product, with special emphasis on human-product interaction.

2) The same intervention but implemented by a therapist via Zoom, Skype, or Teams to continue ensuring protection measures for both the therapist and the patient.

The subjective measures will include the following Psychometric instruments:

1. Post-traumatic diagnostic scale
2. Plutchik Suicide Risk Scale
3. Generalized Anxiety Scale.
4. The Center for Epidemiological Studies Depression Scale-Revised
5. Professional Quality of Life Measure
6. Pittsburgh Sleep Quality Index
7. Scale for measuring resilience with Mexicans
8. Appraisal of Self-care Agency
9. The Fear of COVID-19 Scale
10. Opinion on the treatment.
11. System usability scale

ELIGIBILITY:
Inclusion Criteria:

* To have access to a communication device with access to the internet (computer, tablet, and mobile)
* To have a valid email address.
* To have basic digital skills in the use of an operational system and internet browsing.
* To understand Spanish since all the contents are in this language.
* Symptoms of anxiety, depression, burnout, and fatigue compassion

Exclusion Criteria:

* To have a diagnosis of psychotic disorder
* To be receiving psychological and/or pharmacological treatment during the study
* Moderate to a high score on the suicide scale
* Recent attempt of suicide (3 months)
* To refuse to accept to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-07-16 (Actual); Primary Completion 2022-06-20 (Estimated); Study Completion 2022-06-20 (Estimated)

PRIMARY OUTCOMES:
The Center for Epidemiologic Studies Depression Scale-Revised (CESD-R) | Time Frame: 1 to 1.5 months, depending on the development of the patient and the completion of the 9 nuclear modules.
  The CESD-R is an updated version of the CES-D. The CESD-R consists of 20. This scale assesses the number of depression symptoms within 2 weeks. The scale consists 20 items and contains 4-point score responses (0 to 3) as the following; rarely or none of the time (less than 1 day); some of a little of the time (1-2 days); occasionally or moderate amount of time (3-4 days) and most or all of the time (5-7 days). The total possible range of scores is from 0 to 60 where ^16 is the cut-off point for this scale, and higher scores indicate more symptoms of depression. It is expected a statistically significant decrease (P < 0.05) in depression symptoms.
Decrease in the symptoms of General Anxiety Disorder (GAD-7) | Time Frame: 1 to 1.5 months, depending on the development of the patient and the completion of the 9 nuclear modules.
  On the Generalized Anxiety Disorder 7-item (GAD-7) scale subjects are asked how often, during the last 2 weeks, they have been bothered by each of the 7 core symptoms of generalized anxiety disorder. Response options are "not at all," "several days," "more than half the days," and "nearly every day," scored as 0, 1, 2, and 3, respectively. Therefore, GAD-7 scores range from 0 to 21, with scores of ≥5, ≥10, and ≥15 represent mild, moderate, and severe anxiety symptom levels, respectively. Is expected a statistically significant decrease (P < 0.05) in the General Anxiety symptoms.
Decrease in the score of The Pittsburgh Sleep Quality Index (PSQI). | Time Frame: 1 to 1.5 months, depending on the development of the patient and the completion of the 9 nuclear modules.
  This instrument assesses the quality patterns of sleep. It differentiates the "poor" and "good" sleep by measuring seven areas, where the range score of answers are from 0 to 3, the global sum of this scale can be a value between 0 to 60, and the cutoff point is "5" that indicates a "poor" sleep quality. It is expected a statistically significant decrease (P < 0.05) in the Sleep Quality measure.
Decrease in the scores of the Post-Traumatic Stress Disorder Symptom Scale (PSS) | Time Frame: 1 to 1.5 months, depending on the development of the patient and the completion of the 9 nuclear modules.
  The Post-Traumatic Stress Disorder Symptom Scale is a 17-item structured interview. The severity over the last 2 weeks of each item on the PSS is rated by the interviewer using a 4-point scale: 0 = not at all, 1 = a little bit, 2 = somewhat, and 3 = very much. The maximum possible score is 51 (severely affected) and the minimum possible score is 0 (total absence of the symptoms). The total severity score is calculated as the sum of the severity ratings for the 17 items. The diagnosis of the Post-Traumatic Stress Disorder Symptom Scale is made when at least 1 re-experiencing, 3 avoidance, and 2 arousal symptoms are endorsed on the scale by individuals who were traumatized at least one month prior to the assessment. It is expected a statistically significant decrease (P < 0.05) in the symptoms of Post-Traumatic Stress Disorder in the patients suffering from this disorder.
Increase in the score of the Professional Quality of Life Measure (ProQOL) | Time Frame: 1 to 1.5 months, depending on the development of the patient and the completion of the 9 nuclear modules.
  The professional quality of life will be evaluated with the ProQOL scale (Professional Quality of Life Measure). This scale measures the sections of Satisfaction by empathy, compassion fatigue, and Burnout. The scale is composed of 30 Likert-type questions with five possible answers, being: Never = 1, Rarely = 2, Sometimes = 3, Often = 4 and Often = 5. A score of 17 could indicate affect action in the measured dimensions. It is expected a statistically significant decrease (P < 0.05) in the perception of Professional Quality of Life of the patients.
Increase in the score of the Appraisal of Self-care Agency (ASA) | Time Frame: 1 to 1.5 months, depending on the development of the patient and the completion of the 9 nuclear modules.
  This scale is made up of 24 Likert-type reagents with four types of response, which have a score of one to four points, which when performing the final sum may result in the range of 24-96. The higher the resulting score, the greater the person's self-care capabilities. Maximum ability of self-care is reflected with a score of 96 and a minimum with 24, where high scores of self-care are with scores equal or higher to 76, for a medium ability with equal or higher to 70 but equal or lower than 75 and a low ability any score of 69 or lower. It is expected a statistically significant increase (P < 0.05) in the in the score of the Appraisal of Self-care Agency.

SECONDARY OUTCOMES:
Decrease in the Plutchik Suicide Risk Scale (BSI) | Time Frame: 1 to 1.5 months, depending on the development of the patient and the completion of the 9 nuclear modules.
  The Plutchik Suicide Risk Scale is a structured self-report questionnaire for evaluating Suicide Risk. It consists of 15 items that assess the history of suicide attempts, ideation, and suicide plans. It differentiates patients with a suicide risk from the non-suicide risk. This scale has dichotomous responses of Yes/No, and has a cut-off point of 6, where a point above the cut-off means a higher suicide risk. In this study, the suicidal patients are not considering the depression treatment although is necessary to assess depressive patients to refer to specialized treatment.
Increase in the Scale for measuring resilience with Mexicans (RESI-M) | Time Frame: 1 to 1.5 months, depending on the development of the patient and the completion of the 9 nuclear modules.
  The RESI-M scale is composed of 43 items, the responses are Likert type (totally disagree, disagree, agree, and totally agree). It is expected a statistically significant increase (P < 0.05) in the in the score of resilience

CONTACTS AND LOCATIONS:
Overall Officials: Anabel de la Rosa Gómez, PhD, Study Chair — Universidad Nacional Autonoma de Mexico; Paulina Erika Herdoiza Arroyo, PhD, Study Chair — Universidad Internacional del Ecuador; Rosa Olimpia Castellanos Vargas, MD, Study Chair — Universidad Autonoma de Ciudad Juarez; Joaquín Mateu Molla, PhD, Study Chair — Valencian International University; Luis Farfallini, PhD, Study Chair — University of Buenos Aires; Eduardo Bautista Valerio, BD, Study Chair — Universidad Nacional Autonoma de Mexico
Locations (3):
- Mexico (3):
  - Universidad Autónoma de Ciudad Juárez, Juárez, Chihuahua
  - Universidad de Guadalajara, Guadalajara, Jalisco
  - Universidad Nacional Autónoma de México, México

IPD SHARING:
Plan to Share IPD: Yes
The information will be available in a private server or in a server of the journal(s) that we will publish the articles that will be the result of this study. The protocol of the study is currently in progress to be published, in this article will be included such study protocol, the informed consent is already shared in the register of clinical trials.
Supporting Information: Study Protocol, ICF
Time Frame: This data will be available approximately in June 2022 and it will be permanently available. It will be shared in the databases of the journal where the article(s) will be published.
Access Criteria: Through the servers of the journal(s) where we will publish the articles.

REFERENCES:
- [Background] Lai J, Ma S, Wang Y, Cai Z, Hu J, Wei N, Wu J, Du H, Chen T, Li R, Tan H, Kang L, Yao L, Huang M, Wang H, Wang G, Liu Z, Hu S. Factors Associated With Mental Health Outcomes Among Health Care Workers Exposed to Coronavirus Disease 2019. JAMA Netw Open. 2020 Mar 2;3(3):e203976. doi: 10.1001/jamanetworkopen.2020.3976. PMID 32202646
- [Background] Shechter A, Diaz F, Moise N, Anstey DE, Ye S, Agarwal S, Birk JL, Brodie D, Cannone DE, Chang B, Claassen J, Cornelius T, Derby L, Dong M, Givens RC, Hochman B, Homma S, Kronish IM, Lee SAJ, Manzano W, Mayer LES, McMurry CL, Moitra V, Pham P, Rabbani L, Rivera RR, Schwartz A, Schwartz JE, Shapiro PA, Shaw K, Sullivan AM, Vose C, Wasson L, Edmondson D, Abdalla M. Psychological distress, coping behaviors, and preferences for support among New York healthcare workers during the COVID-19 pandemic. Gen Hosp Psychiatry. 2020 Sep-Oct;66:1-8. doi: 10.1016/j.genhosppsych.2020.06.007. Epub 2020 Jun 16. PMID 32590254
- [Background] Paul V, Patel S, Royse M, Odish M, Malhotra A, Koenig S. Proning in Non-Intubated (PINI) in Times of COVID-19: Case Series and a Review. J Intensive Care Med. 2020 Aug;35(8):818-824. doi: 10.1177/0885066620934801. PMID 32633215
- [Background] Allan SM, Bealey R, Birch J, Cushing T, Parke S, Sergi G, Bloomfield M, Meiser-Stedman R. The prevalence of common and stress-related mental health disorders in healthcare workers based in pandemic-affected hospitals: a rapid systematic review and meta-analysis. Eur J Psychotraumatol. 2020 Oct 16;11(1):1810903. doi: 10.1080/20008198.2020.1810903. PMID 33244359
- [Background] Pappa S, Ntella V, Giannakas T, Giannakoulis VG, Papoutsi E, Katsaounou P. Prevalence of depression, anxiety, and insomnia among healthcare workers during the COVID-19 pandemic: A systematic review and meta-analysis. Brain Behav Immun. 2020 Aug;88:901-907. doi: 10.1016/j.bbi.2020.05.026. Epub 2020 May 8. PMID 32437915
- [Background] Luo M, Guo L, Yu M, Jiang W, Wang H. The psychological and mental impact of coronavirus disease 2019 (COVID-19) on medical staff and general public - A systematic review and meta-analysis. Psychiatry Res. 2020 Sep;291:113190. doi: 10.1016/j.psychres.2020.113190. Epub 2020 Jun 7. PMID 32563745
- [Background] Smith GD, Ng F, Ho Cheung Li W. COVID-19: Emerging compassion, courage and resilience in the face of misinformation and adversity. J Clin Nurs. 2020 May;29(9-10):1425-1428. doi: 10.1111/jocn.15231. Epub 2020 Mar 10. No abstract available. PMID 32155302
- [Background] Hossain F, Clatty A. Self-care strategies in response to nurses' moral injury during COVID-19 pandemic. Nurs Ethics. 2021 Feb;28(1):23-32. doi: 10.1177/0969733020961825. Epub 2020 Oct 30. PMID 33124492
- [Background] Williamson V, Stevelink SAM, Greenberg N. Occupational moral injury and mental health: systematic review and meta-analysis. Br J Psychiatry. 2018 Jun;212(6):339-346. doi: 10.1192/bjp.2018.55. PMID 29786495
- [Background] Drissi N, Ouhbi S, Marques G, de la Torre Diez I, Ghogho M, Janati Idrissi MA. A Systematic Literature Review on e-Mental Health Solutions to Assist Health Care Workers During COVID-19. Telemed J E Health. 2021 Jun;27(6):594-602. doi: 10.1089/tmj.2020.0287. Epub 2020 Sep 22. PMID 32970532
- [Background] Yang L, Yin J, Wang D, Rahman A, Li X. Urgent need to develop evidence-based self-help interventions for mental health of healthcare workers in COVID-19 pandemic. Psychol Med. 2021 Jul;51(10):1775-1776. doi: 10.1017/S0033291720001385. Epub 2020 Apr 28. No abstract available. PMID 32340642
- [Background] Koslowsky M, Bleich A, Greenspoon A, Wagner B, Apter A, Solomon Z. Assessing the validity of the Plutchik Suicide Risk Scale. J Psychiatr Res. 1991;25(4):155-8. doi: 10.1016/0022-3956(91)90019-7. PMID 1779413
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Result] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Result] Novy DM, Stanley MA, Averill P, Daza P. Psychometric comparability of English- and Spanish-language measures of anxiety and related affective symptoms. Psychol Assess. 2001 Sep;13(3):347-55. doi: 10.1037//1040-3590.13.3.347. PMID 11556271
- [Result] Foa EB, Cashman L, Jaycox L, Perry K. The validation of a self-report measure of posttraumatic stress disorder: the Posttraumatic Diagnostic Scale. Psychological assessment. 1997 Dec;9(4):445.
- [Result] González-Forteza C, Torres CS, Tapia AJ, Fernández IH, González-González A, Garcia FJ, Medina-Mora ME, Mejía HFV. Confiabilidad y validez de la escala de depresión CES-D en un censo de estudiantes de nivel medio superior y superior, en la Ciudad de México [Reliability and validity of the depression scale CES-D in high school and college students from Mexico City: Results from a census]. Salud Mental. 2011; 34(1): 53-59.
- [Result] Garcia-Campayo J, Zamorano E, Ruiz MA, Pardo A, Perez-Paramo M, Lopez-Gomez V, Freire O, Rejas J. Cultural adaptation into Spanish of the generalized anxiety disorder-7 (GAD-7) scale as a screening tool. Health Qual Life Outcomes. 2010 Jan 20;8:8. doi: 10.1186/1477-7525-8-8. PMID 20089179
- [Result] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Result] Ahorsu DK, Lin CY, Imani V, Saffari M, Griffiths MD, Pakpour AH. The Fear of COVID-19 Scale: Development and Initial Validation. Int J Ment Health Addict. 2022;20(3):1537-1545. doi: 10.1007/s11469-020-00270-8. Epub 2020 Mar 27. PMID 32226353
- [Result] Healy DJ, Barry K, Blow F, Welsh D, Milner KK. Routine use of the Beck Scale for Suicide Ideation in a psychiatric emergency department. Gen Hosp Psychiatry. 2006 Jul-Aug;28(4):323-9. doi: 10.1016/j.genhosppsych.2006.04.003. PMID 16814632
- [Derived] Dominguez-Rodriguez A, Martinez-Arriaga RJ, Herdoiza-Arroyo PE, Bautista-Valerio E, de la Rosa-Gomez A, Castellanos Vargas RO, Lacomba-Trejo L, Mateu-Molla J, Lupercio Ramirez MJ, Figueroa Gonzalez JA, Ramirez Martinez FR. E-Health Psychological Intervention for COVID-19 Healthcare Workers: Protocol for its Implementation and Evaluation. Int J Environ Res Public Health. 2022 Oct 5;19(19):12749. doi: 10.3390/ijerph191912749. PMID 36232049

DOCUMENTS (1):
  • Informed Consent Form (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/65/NCT04890665/ICF_000.pdf